CLINICAL TRIAL: NCT06365294
Title: Rescue Extracranial Vertebral Stenting in Tandem Occlusions
Acronym: REVET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Cuong Tran Chi (Other)
Responsible Party: Sponsor-Investigator, Dr. Cuong Tran Chi, Director - Doctor, Can Tho Stroke International Services Hospital
Organization: Can Tho Stroke International Services Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REVET Study
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Acute Stroke; Ischemic Stroke, Acute; Vertebro Basilar Ischemia
Keywords: tandem occlusions; posterior circulation; rescue extracrnial stenting
MeSH Terms: conditions — Stroke; Ischemic Stroke; Vertebrobasilar Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rescue extracranial vertebral stenting (Experimental): Rescue extracranial vertebral stenting in tandem occlusions
  Interventions: Procedure: Rescue extracranial stenting

INTERVENTIONS:
Procedure: Rescue extracranial stenting — Rescue extracranial stenting in tandem occlusions

SUMMARY:
The acute vertebrobasilar occlusion associated with the poor prognosis, particularly tandem occlusion. However, few data on the efficacy of the endovascular therapy was indicated in this occlusion. The investigators reported whether the additional rescue extracranial stenting improved clinical outcome by modified Rankin Scale (mRS) score within 3 months after the procedure

DETAILED DESCRIPTION:
Acute vertebrobasilar artery occlusion is one of the cerebrovascular diseases with high disability and mortality rates. Although mechanical thrombectomy has recently been demonstrated an effective treatment for large vessel occlusions of posterior circulation, the treatment strategies depending on the specific pathophysiology. Tandem occlusion in posterior circulation is less frequently than in anterior one, comprises severe stenosis or occlusion of the extracranial vertebral artery ipsilateral to its intracranial and basilar occlusion. The recent studies showed the benefit of the "distal-to-proximal" approach, there were many tecniques to achieved the successful recanalization. Besides, the use of Dotter technique allowed 8F guiding catheter to cross the extracranial lesions easily and save the procedural time. However, the Diagnosis 5F-Dotter, like the Dilator-Dotter, has not been mentioned in previous studies. Therefore, the aim of the our study was to assess the improvement of outcomes at 3 months posttreatment in patients receiving rescue extracranial vertebral stenting

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Onset to treatment time < 24 hours
* NIHSS > 5
* pc-ASPECTS ≥ 5

Exclusion Criteria:

* Premorbid mRS > 2
* Extensive, bilateral brain-stem infarction on neuroimaging
* Cerebellar mass effect on neuroimaging
* Loss to follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
The good 3-month outcome rate | 3 months
  The good 3-month outcome rate was accessed by modified Rankin Score (mRS ≤ 2).

CONTACTS AND LOCATIONS:
Overall Officials: Can Tho Stroke International Services Hospital, Study Director — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho SIS Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen JE, Leker RR, Gomori JM, Eichel R, Rajz G, Moscovici S, Itshayek E. Emergent revascularization of acute tandem vertebrobasilar occlusions: Endovascular approaches and technical considerations-Confirming the role of vertebral artery ostium stenosis as a cause of vertebrobasilar stroke. J Clin Neurosci. 2016 Dec;34:70-76. doi: 10.1016/j.jocn.2016.05.005. Epub 2016 Aug 10. PMID 27522497
- [Background] Han N, Ma L, Zhao L, Xu G, Jia Y, Wang H. The Dilator-Dotter technique can successfully treat tandem lesions of posterior circulation. Medicine (Baltimore). 2024 Jan 26;103(4):e37044. doi: 10.1097/MD.0000000000037044. PMID 38277540